CLINICAL TRIAL: NCT06880198
Title: An Interventional, Not Pharmacological Study to Evaluate Impact® as Support to Anti PD1 or Anti PD1 Based Regimen Treatment in Patients With Inoperable Locally Advanced or Metastatic Melanoma
Brief Title: Study to Evaluate Impact® as Support to Anti PD1 or Anti PD1 Based Regimen Treatment in Patients With Inoperable Locally Advanced or Metastatic Melanoma
Acronym: MELA-IMPACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Melanoma Onlus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MELA-IMPACT
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Melanoma Metastatic; Locally Advanced Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oral Impact®: single arm (Experimental): The patients will be treated with Oral Impact® administered at the dose of two bricks/day for 21 days + one brick/day for 14 days, starting exactly one week before Anti PD-1 treatment (nivolumab) or anti PD1 based regimen therapy (Nivolumab plus Ipilimumab or Nivolumab plus Relatlimab)as per clinical practice, administered up to two years.
  Interventions: Dietary Supplement: Oral Impact®

INTERVENTIONS:
Dietary Supplement: Oral Impact® — One Arm: 2 Impact brick/d for 21 days + 1 brick/d for 14 days, starting exactly one week before Anti PD-1 treatment in patients with inoperable locally advanced or metastatic melanoma Treatment duration: 35 days

SUMMARY:
This is a monocentric, prospective study evaluating the effectiveness in reducing immune-related adverse events, and translational study conducted on 20 patients with inoperable locally advanced or metastatic melanoma.

The patients will be treated with Oral Impact® administered at the dose of two bricks/day for 21 days + one brick/day for 14 days, starting exactly one week before Anti PD-1 treatment (nivolumab) or anti PD1 based regimen therapy (Nivolumab plus Ipilimumab or Nivolumab plus Relatlimab) as per clinical practice.

The comparison will be done with historical literature data on patients matched by age, sex, disease stage, and therapy dosage, not treated with Impact.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Histologically confirmed stage III (unresectable) or stage IV Cutaneous Melanoma;
3. PD-L1 evaluation and as per standard clinical practice, patients with PD-L1 < 1% will be treated with anti PD1 based regimen and patients with PD-L1>1% will be treated with anti-PD1 in monotherapy;
4. Anti-PD1 (Nivolumab) or anti PD1 based regimen (Nivolumab plus Ipilimumab or Nivolumab plus Relatlimab) planned as per standard clinical practice and decision by the treating oncologist; ;
5. Measurable disease by computed tomography (CT) or Magnetic Resonance Imaging (MRI) per RECIST 1.1 criteria;
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1;
7. Screening laboratory values must meet the following criteria before starting the treatment:

   1. WBCs ≥2000/μL
   2. Neutrophils ≥1500/μL
   3. Platelets ≥100 x 10³/μL
   4. Hemoglobin ≥9.0 g/dL
   5. Serum creatinine of ≤1.5 times the upper normal limits or creatinine clearance >40 mL/minute
   6. AST ≤ 3 times the upper normal limits
   7. ALT ≤ 3 times the upper normal limits
   8. Total bilirubin ≤1.5 times the upper normal limits (except patients with Gilbert Syndrome who must have total bilirubin <3.0 mg/dL)
8. Prior palliative radiotherapy must have been completed at least 2 weeks prior to study drug administration;
9. Patients of reproductive potential, must use adequate contraception methods;
10. Signed written consent form;

Exclusion Criteria:

1. Active brain metastases;
2. Patients with previous malignancies unless a complete remission was achieved at least 2 years prior to study entry;
3. Patients with prior systemic anticancer therapy for unresectable or metastatic melanoma;
4. Any serious or uncontrolled medical disorder or active infection that, in the opinion of the investigator, may increase the risk associated with study participation, study drug administration, or would impair the ability of the patient to receive protocol therapy;
5. Presence of active, known, or suspected autoimmune disease;
6. Subjects with a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days of treatment;
7. Participation in any interventional drug or medical device study within 30 days prior to treatment start;
8. Patients with active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or active C hepatitis or active HIV;
9. History of severe hypersensitivity reactions to other monoclonal antibodies;
10. Pregnant and breast-feeding women;
11. Patients of reproductive who refuse to use effective methods of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
the role of immunonutrition with Oral Impact® in reducing G3 - G4 irAEs frequency and severity grade of anti-PD1 therapy (Nivolumab) or anti-PD1 based regimen in patients with inoperable locally advanced or metastatic melanoma. | up to 12 months from EoT

SECONDARY OUTCOMES:
Prognostic bio-markers evaluation | from day -7 up to EoT
  Evaluation of peripheral blood biomarkers, metagenomic sequencing of gut microbiota, gene profile analysis, and, if archived tissues are available, tumor tissue biomarkers.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Nazionale Tumori IRCCS - Fondazione "G. Pascale", Napoli, Italy

IPD SHARING:
Plan to Share IPD: No